CLINICAL TRIAL: NCT04449640
Title: Uterine Rupture in Pregnancy After Hysteroscopic Septum Resection: a Twenty-year Retrospective Analysis
Brief Title: Uterine Rupture After Hysteroscopic Septum Resection
Status: Completed | Type: Observational
Sponsor: Università degli Studi dell'Insubria (Other)
Collaborators: University of Ljubljana (Other); Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Antonio Simone Laganà, Principal Investigator, Università degli Studi dell'Insubria
Other Study IDs: URAHSR-1
Record Dates: First submitted 2020-06-24; First posted 2020-06-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Septum; Uterus; Rupture, Uterine
Keywords: Hysteroscopy; Uterine septum; Complications; Uterine perforation; Pregnancy; Uterine rupture
MeSH Terms: conditions — Uterine Rupture; Septate Uterus; Uterine Perforation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Uterine rupture: Women who had uterine rupture during pregnancy.
  Interventions: Procedure: Hysteroscopic septum resection.

INTERVENTIONS:
Procedure: Hysteroscopic septum resection. — Resection of a uterine septum by hysteroscopic surgery.

SUMMARY:
To date, several studies have already confirmed a positive effect of hysteroscopic metroplasty on reproductive outcomes in primary infertile women affected by uterine septum, the most common uterine malformation. Nevertheless, very few data are available about the risk of uterine rupture in subsequent pregnancies after hysteroscopic septum resection (HSR). In order to shed about this element, we will retrospectively review the cases of uterine rupture in our setting in the last twenty years, identify which of them had previously undergone HSR, and evaluate the main clinical characteristics for each case.

ELIGIBILITY:
Inclusion Criteria:

* Previous hysteroscopic septum resection;
* Pregnancy;
* Uterine rupture.

Exclusion Criteria:

* Previous myomectomy (regardless of the surgical technique) or cesarean section.

Ages: 18 Years to 48 Years | Sex: Female
Age Groups: Adult
Study Population: Pregnant women who underwent previous hysteroscopic septum resection.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Uterine rupture | Retrospective analysis over the last twenty years.
  Rupture of muscular wall of the uterus tears during pregnancy or childbirth.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Simone Laganà, M.D., Ph.D., Study Chair — Università degli Studi dell'Insubria; Helena Ban Frangež, M.D., Ph.D., Study Director — University of Ljubljana
Locations (1):
- Antonio Simone Laganà, Ljubljana, Italy

IPD SHARING:
Plan to Share IPD: Undecided